CLINICAL TRIAL: NCT05421156
Title: Evaluation of Long-term Sexual Dysfunctions, Urinary Dysfunctions and Pelvic Organ Prolapse in Women Who Underwent Laparoscopic Subtotal Versus Total Hysterectomy for Benign Conditions
Brief Title: Long-term Outcomes After Laparoscopic Subtotal and Total Hysterectomy
Acronym: LAST-1
Status: Not yet recruiting | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, University of Palermo
Other Study IDs: LAST-1
Record Dates: First submitted 2022-06-12; First posted 2022-06-16 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Hysterectomy
Keywords: Subtotal Laparoscopic Hysterectomy; Total Laparoscopic Hysterectomy; Hysterectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subtotal Laparoscopic Hysterectomy: Women who underwent subtotal laparoscopic hysterectomy
  Interventions: Procedure: Subtotal Laparoscopic Hysterectomy
- Total Laparoscopic Hysterectomy: Women who underwent total laparoscopic hysterectomy
  Interventions: Procedure: Total Laparoscopic Hysterectomy

INTERVENTIONS:
Procedure: Subtotal Laparoscopic Hysterectomy — Subtotal laparoscopic hysterectomy involves removing the main body of the uterus and leaving the cervix in place by laparoscopy.
  Groups: Subtotal Laparoscopic Hysterectomy
Procedure: Total Laparoscopic Hysterectomy — Total laparoscopic hysterectomy involves removing the whole uterus and cervix by laparoscopy
  Groups: Total Laparoscopic Hysterectomy

SUMMARY:
Hysterectomy is one of the most commonly performed gynecologic surgeries in the USA. It is used for many benign conditions such as leiomyoma and abnormal uterine bleeding. Surgery may involve the removal of the cervix (total hysterectomy, TH) or its preservation (supracervical or subtotal hysterectomy, SH). Whether TH or SH is the best procedure for benign conditions is a matter of debate. Considering the lack of evidence, this study aims to evaluate long-term sexual dysfunctions, urinary dysfunctions and pelvic organ prolapse in women who underwent laparoscopic subtotal versus total hysterectomy for benign conditions.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent subtotal or total hysterectomy by laparoscopy for benign conditions.

Exclusion Criteria:

* Women with gynecological and non-gynecological cancers.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who underwent subtotal or total hysterectomy by laparoscopy for benign conditions
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Sexual Dysfunctions | 5 years after surgery
  Female Sexual Function Index

SECONDARY OUTCOMES:
Urinary Dysfunctions | 5 years after surgery
  Pelvic Floor Distress Inventory short form
Pelvic Organ Prolapse | 5 years after surgery
  Pelvic Organ Prolapse (POP-Q) evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Ph.D., Principal Investigator — University of Palermo

IPD SHARING:
Plan to Share IPD: Undecided